CLINICAL TRIAL: NCT05581303
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study Assessing the Impact of Olpasiran on Major Cardiovascular Events in Participants With Atherosclerotic Cardiovascular Disease and Elevated Lipoprotein(a)
Brief Title: Olpasiran Trials of Cardiovascular Events and Lipoprotein(a) Reduction (OCEAN(a)) - Outcomes Trial
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20180244
Expanded Access: NCT07079267 (Available)
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: Atherosclerotic Cardiovascular Disease; ASCVD; AMG 890; Olpasiran
MeSH Terms: conditions — Atherosclerosis | interventions — olpasiran

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo will be administered by subcutaneous injection
  Interventions: Drug: Placebo
- Olpasiran (Experimental): Olpasiran will be administered by subcutaneous injection
  Interventions: Drug: Olpasiran

INTERVENTIONS:
Drug: Placebo — Placebo given by subcutaneous injection once every 12 weeks (Q12W).
  Arms: Placebo
Drug: Olpasiran — Olpasiran given by subcutaneous injection Q12W.
  Arms: Olpasiran

SUMMARY:
The primary objective of this study is to compare the effect of treatment with olpasiran, to placebo, on the risk for coronary heart disease death (CHD death), myocardial infarction, or urgent coronary revascularization in participants with atherosclerotic cardiovascular disease (ASCVD) and elevated Lipoprotein(a).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to ≤ 85 years
* Lp(a)≥ 200 nmol/L during screening
* History of ASCVD as evidenced by history of either:

  * Myocardial infarction (presumed type 1 event due to plaque rupture/erosion) and/or
  * Coronary revascularization with percutaneous coronary intervention AND at least 1 additional risk factor.

Exclusion Criteria:

* Severe renal dysfunction
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN), or total bilirubin (TBL) > 2 x ULN during screening
* History of hemorrhagic stroke
* History of major bleeding disorder
* Planned cardiac surgery or arterial revascularization
* Severe heart failure
* Current, recent, or planned lipoprotein apheresis
* Previously received ribonucleic acid therapy specifically targeting Lp(a)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7297 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2026-12-29 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
Time to CHD death, myocardial infarction, or urgent coronary revascularization, whichever occurs first | Approximately 4 years

SECONDARY OUTCOMES:
Time to cardiovascular death, myocardial infarction, or ischemic stroke, whichever occurs first | Approximately 4 years
Time to cardiovascular death, myocardial infarction, urgent coronary revascularization, or ischemic stroke, whichever occurs first | Approximately 4 years
Percent change from baseline to Week 48 in Lipoprotein(a) | Baseline and Week 48
Time to myocardial infarction | Approximately 4 years
Time to CHD death or myocardial infarction, whichever occurs first | Approximately 4 years
Time to urgent coronary revascularization | Approximately 4 years
Time to coronary revascularization | Approximately 4 years
Time to CHD death | Approximately 4 years
Time to cardiovascular death | Approximately 4 years
Time to death by any cause | Approximately 4 years
Time to ischemic stroke | Approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (737):
- United States (133):
  - Ascension Saint Vincents Birmingham, Birmingham, Alabama
  - Grandview Medical Center Affinity Cardiovascular Specialists, LLC, Birmingham, Alabama
  - Heart Center Research LLC, Huntsville, Alabama
  - Mobile Heart Specialists PC, Mobile, Alabama
  - Alaska Cardiovascular Research Foundation, Anchorage, Alaska
  - Elite Clinical Studies LLC, Phoenix, Arizona
  - HonorHealth Research and Innovation Institute, Scottsdale, Arizona
  - National Heart Institute, Beverly Hills, California
  - Vitality Clinical Research, Beverly Hills, California
  - University of California San Diego, La Jolla, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of California Irvine, Orange, California
  - University of California Los Angeles, Santa Monica, California
  - Manshadi Heart Institute, Stockton, California
  - Med Partners, Inc dba Premiere Medical Center, Inc, Toluca Lake, California
  - UCHealth Memorial Central, Colorado Springs, Colorado
  - Cardiology Associates of Fairfield County PC, Stamford, Connecticut
  - MedStar Clinical Research, Washington D.C., District of Columbia
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Bay Area Cardiology, Brandon, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Cardiology Associates Research LLC, Daytona Beach, Florida
  - Jellinger and Lerman MD PA dba The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - Elite Cardiac Research Center LLC, Hialeah, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - University of Florida, Jacksonville, Florida
  - East Coast Institute for Research LLC, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Advanced Research for Health Improvement, LLC, Naples, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - AdventHealth Medical Group Cardiology at Orlando, Orlando, Florida
  - East Coast Institute for Research, LLC, Saint Augustine, Florida
  - Saint Johns Center for Clinical Research, Saint Augustine, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Care Access - Tampa, Tampa, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Morehouse School of Medicine, Atlanta, Georgia
  - Northeast Georgia Medical Center Wisteria Building, Cumming, Georgia
  - NSC Research, Johns Creek, Georgia
  - St Lukes Idaho Cardiology Associates, Meridian, Idaho
  - Northwest Heart Clinical Research LLC, Arlington Heights, Illinois
  - Northshore University Health System, Evanston, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Cardiovascular Research of Northwest Indiana LLC, Munster, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - MercyOne Iowa Heart Center, West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Midwest Heart and Vascular Specialists, Overland Park, Kansas
  - Saint Elizabeth Covington, Covington, Kentucky
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - University of Louisville Health - Jewish Hospital, Louisville, Kentucky
  - Louisiana Heart Center, Hammond, Louisiana
  - Care Access - Lake Charles, Lake Charles, Louisiana
  - Clinical Trials of America Inc, Monroe, Louisiana
  - Monroe Research LLC, West Monroe, Louisiana
  - Northern Light Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Metropolitan Cardiovascular Consultants LLC, Beltsville, Maryland
  - TidalHealth Peninsula Regional, Inc, Salisbury, Maryland
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Advanced Cardiology Associates, Grand Rapids, Michigan
  - Healthy Heart Cardiology, Grand Rapids, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Arcturus Healthcare, Public Limited Company, Troy Internal Medicine Research Division, Troy, Michigan
  - Fairview Health Services, Maplewood, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Cardiology Associates Research LLC, Tupelo, Mississippi
  - Saint Louis Heart and Vascular PC, St Louis, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - Palm Research Center Inc, Las Vegas, Nevada
  - Renown Institute for Heart and Vascular Health, Reno, Nevada
  - Saint Michaels Medical Center, Newark, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - New York Presbyterian Medical Group Hudson Valley Cardiology, Cortlandt Manor, New York
  - Elligo Health Research, Kew Gardens, New York
  - WMCHealth Heart and Vascular Institute Kingston Division of Cardiology, Kingston, New York
  - Northwell Health Physician Partners Cardiology at Manhasset, Manhasset, New York
  - New York University Langone Health, New York, New York
  - Northwell Health Lenox Hill Heart and Vascular, New York, New York
  - Icahn School of Medicine at Mount Sinai Queens, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Northwell Health Physician Partners at Peconic, Riverhead, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Westchester Medical Center, Valhalla, New York
  - NY Family Docs, Woodhaven, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Moses H Cone Memorial Hospital, Greensboro, North Carolina
  - Lapis Clinical Research, Mooresville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - TriHealth Good Samaritan Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The OhioHealth Research Institute, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Rama Research LLC, Marion, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Capital Area Research LLC, Newport, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Montefiore Medical Center - Bronx, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Midlands Cardiology, Columbia, South Carolina
  - Piedmont Research Partners, Fort Mill, South Carolina
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Stern Cardiovascular Foundation Inc, Germantown, Tennessee
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Baylor Scott and White Heart and Vascular Hospital-Dallas, Dallas, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - David Turbay, MD, El Paso, Texas
  - Care Access - Georgetown, Georgetown, Texas
  - Baylor College of Medicine, Houston, Texas
  - Texas Cardiology Associates of Houston, Kingwood, Texas
  - Texas Institute of Cardiology, McKinney, Texas
  - Permian Research Foundation, Odessa, Texas
  - Northwest Houston Heart Center, Tomball, Texas
  - Inova Heart and Vascular Institute, Fairfax, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Virginia Heart - Loudoun, Leesburg, Virginia
  - Carient Heart and Vascular, Manassas, Virginia
  - Bon Secours Cardiology, Midlothian, Virginia
  - Tidewater Physicians Multispecialty Group Clinical Research, Newport News, Virginia
  - Winchester Cardiology and Vascular Medicine, Winchester, Virginia
  - Pulse Heart Institute, Puyallup, Washington
- Argentina (25):
  - Instituto de Investigaciones Clinicas Bahia Blanca, Bahía Blanca, Buenos Aires
  - Cedic Centro de Investigacion Clinica, CABA, Buenos Aires
  - Ciprec Centro de Investigacion y Prevencion Cardiovascular, CABA, Buenos Aires
  - Cinme - Centro de Investigaciones Metabolicas, CABA, Buenos Aires
  - Consultorio Medico Dr Litvak Bruno, CABA, Buenos Aires
  - Cemedic Centro de Especialidades Medicas, CABA, Buenos Aires
  - Centro Medico Dra Laura Maffei Investigacion Clinica Aplicada, CABA, Buenos Aires
  - Consultorios Medicos Dr Besada, CABA, Buenos Aires
  - Fundacion Respirar - Consultorios Medicos Dr Doreski, CABA, Buenos Aires
  - Glenny Corp SA, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Fundacion Favaloro, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Icba Instituto Cardiovascular de Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Cuidad Autonoma de Buenos Aires, Buenos Aires
  - Ciad - Consultorio Integral de Atencion al Diabetico, Morón, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes, Buenos Aires
  - Instituto de Investigaciones Clinicas de San Nicolas, San Nicolás de los Arroyos, Buenos Aires
  - Instituto de Investigaciones Clinicas Zarate, Zárate, Buenos Aires
  - Clinica Privada del Prado, Córdoba, Córdoba Province
  - Instituto Latinoamericano de Investigaciones Medicas Cidim-Ilaim, Córdoba, Córdoba Province
  - Instituto de Investigaciones Clinicas de Cordoba, Córdoba, Córdoba Province
  - Clinica Fusavim Privada SRL, Villa María, Córdoba Province
  - Instituto de Investigaciones Clinicas Rosario, Rosario, Santa Fe Province
  - Clinica Adventista Belgrano, Buenos Aires
  - Instituto Medico Damic, Córdoba
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
- Australia (23):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Advara HeartCare Wesley, Auchenflower, Queensland
  - Advara HeartCare Bundaberg, Bundaberg, Queensland
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Core Research Group Pty Ltd, Milton, Queensland
  - Dr Heart Pty Ltd, Woolloongabba, Queensland
  - Nightingale Research, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Advara HeartCare Leabrook, Leabrook, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Advara HeartCare Berwick, Berwick, Victoria
  - Victorian Heart Hospital, Clayton, Victoria
  - The Cardiologists Proprietary Limited, Epping, Victoria
  - Barwon Health Geelong Hospital, Geelong, Victoria
  - Advara HeartCare Ringwood, Ringwood, Victoria
  - Advara HeartCare Joondalup, Joondalup, Western Australia
  - Mount Hospital, Murdoch, Western Australia
  - Linear Clinical Research Limited, Nedlands, Western Australia
- Austria (11):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Medizinische Universitaet Graz, Graz
  - Klinikum Klagenfurt am Woerthersee, Klagenfurt
  - Krankenhaus der Barmherzigen Brueder Linz, Linz
  - Landeskrankenhaus Salzburg, Salzburg
  - Universitaetsklinikum Sankt Poelten, Sankt Pölten
  - Klinik Landstrasse, Vienna
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
  - Klinik Hietzing, Vienna
  - Klinik Ottakring, Vienna
  - Krankenhaus Nord - Klinik Floridsdorf, Vienna
- Belgium (13):
  - Algemeen Stedelijk Ziekenhuis Aalst, Aalst
  - Onze Lieve Vrouw Ziekenhuis - campus Aalst, Aalst
  - Ziekenhuisnetwerk Antwerpen site Cadix, Antwerp
  - Cliniques universitaires de Bruxelles Hopital Erasme, Brussels
  - Algemeen Ziekenhuis Sint Blasius, Dendermonde
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Ziekenhuis Oost-Limburg - Campus Sint-Jan, Genk
  - Algemeen Ziekenhuis Sint Lucas, Ghent
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Regional de la Citadelle, Liège
  - Algemeen Ziekenhuis Sint-Maarten, Mechelen
  - Algemeen Ziekenhuis Turnhout, Turnhout
- Brazil (39):
  - Hospital Universitario Walter Cantidio, Fortaleza, Ceará
  - Centro de Pesquisas em Diabetes e Doencas Endocrino Metabolicas, Fortaleza, Ceará
  - Centro do Diagnostico e Pesquisa da Osteoporose do Espirito Santo, Vitória, Espírito Santo
  - Hospital Santa Izabel, Salvador, Estado de Bahia
  - Hospital Ana Nery, Salvador, Estado de Bahia
  - Instituto de Ensino e Pesquisa do Hospital da Bahia, Salvador, Estado de Bahia
  - Associacao de Amparo a Saude Ensino e Pesquisa, Brasília, Federal District
  - Hospital das Clinicas da Universidade Federal de Goias, Goiânia, Goiás
  - Hospital Universitario Maria Aparecida Pedrossian, Campo Grande, Mato Grosso do Sul
  - Eurolatino Pesquisas Medicas, Uberlândia, Minas Gerais
  - Quanta Diagnostico por Imagem, Curitiba, Paraná
  - Nucleo de Pesquisa Clinica, Curitiba, Paraná
  - Procape, Recife, Pernambuco
  - Hospital Agamenon Magalhaes, Recife, Pernambuco
  - Instituto Atena de Pesquisa Clínica, Natal, Rio Grande do Norte
  - Hospital Sao Francisco da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clínica Associação Hospitalar Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Nucleo de Pesquisa Clinica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Imv Pesquisa Cardiologica, Porto Alegre, Rio Grande do Sul
  - FZ Pesquisa e Servicos em Cardiologia LTDA, Porto Alegre, Rio Grande do Sul
  - AngioCor Blumenau, Blumenau, Santa Catarina
  - jmf Clinica do Coracao ltda, Aracaju, Sergipe
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - Loema Instituto de Pesquisa Clinica e Consultores Ltda, Campinas, São Paulo
  - icm Instituto do Coração de Marilia, Marília, São Paulo
  - Clinicor Clinica Cardiologica Ltda, Ribeirão Preto, São Paulo
  - Hospital Das Clinicas da Faculdade de Medicina de Ribeirao Preto da Universidade de Sao Paulo, Ribeirão Preto, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Instituto de Pesquisa em Endocrinologia Clinica IPEC, São Paulo, São Paulo
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - Instituto do Coracao do Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo
  - Integral Pesquisa e Ensino, Votuporanga, São Paulo
  - IBPClin Instituto Brasil de Pesquisa Clinica, Rio de Janeiro
  - Fundacao Pro-Coracao, Rio de Janeiro
  - Centro Paulista de Investigacoes Clinicas Cepic, São Paulo
- Bulgaria (13):
  - Multiprofile Hospital for Active Treatment Puls AD, Blagoevgrad
  - Multiprofile Hospital for Active Treatment - Haskovo AD, Haskovo
  - Medical Center Medconsult Pleven OOD, Pleven
  - Multiprofile Hospital for Active Treatment Heart and Brain EAD, Pleven
  - Medical Center Cardiomed 2020 EOOD, Sliven
  - Diagnostic-Consultative Center Ascendent OOD, Sofia
  - Multiprofile Hospital for Active Treatment National Hospital of Cardiology EAD, Sofia
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
  - Medical Center Kalimat EOOD, Sofia
  - Medical Centre Synexus Sofia EOOD, Sofia
  - Medical Center Orpheus OOD, Stara Zagora
  - Ambulatory for Individual Practice for Specialized Medical Care - Kardio EOOD, Varna
- Canada (20):
  - ARC Biosystems Incorporated, Vancouver, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - Discovery Clinical Services Ltd, Victoria, British Columbia
  - LMC Clinical Research Incorporated, Brampton, Ontario
  - Brampton Clinical Trials, Brampton, Ontario
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - LMC Clinical Research Incorporated Thornhill, Concord, Ontario
  - Hamilton Health Sciences Hamilton General Hospital, Hamilton, Ontario
  - One Heart Care, Mississauga, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Oakville Cardiovascular Research, Oakville, Ontario
  - Womens College Hospital, Toronto, Ontario
  - CPS Research, Waterloo, Ontario
  - Ecogene-21 Research, Chicoutimi, Quebec
  - Institut de recherches cliniques de Montreal, Montreal, Quebec
  - Research Institute of McGill University Health Center - Glen Site, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Centre Hotel-Dieu de Quebec, Québec, Quebec
  - Institut Universitaire de cardiologie et de pneumologie de Quebec, Québec, Quebec
  - Clinique des Maladies Lipidiques de Quebec Incorporated, Québec, Quebec
  - Centre de sante et de services sociaux du Nord de Lanaudiere, Saint-Charles-Borromée, Quebec
- China (43):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital ,Sun-Yat Sen University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Huizhou Central Peoples Hospital, Huizhou, Guangdong
  - The Peoples Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Second Nanning Peoples Hospital, Nanning, Guangxi
  - Daqing Oilfield general Hospital, Daqing, Heilongjiang
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Nanyang Second General Hospital, Nanyang, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi Peoples Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The Second Affiliated Hospital to Nanchang University, Nanchang, Jiangxi
  - Jilin Province Peoples Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The Peoples Hospital of Liaoning Province, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shaanxi Provincial Peoples Hospital, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Peoples Hospital, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Zhejiang Provincial Peoples Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Qingdao Fuwai Cardiovascular Hospital, Qingdao
  - Shanghai General Hospital, Shanghai
  - Shanghai Yangpu District Central Hospital（ Yangpu Hospital Affiliated to Tongji University）, Shanghai
  - Renmin Hospital of Wuhan University, Wuhan
  - Zhejiang Hospital, Zhejiang
- Czechia (38):
  - Jessenia as, Nemocnice Beroun, Beroun
  - Hornicka nemocnice s poliklinikou spol sro, Bílina
  - Medicus Services sro, Brandýs nad Labem
  - MTE Medical Center, Brno
  - Centrum pro zdravi sro, Brno
  - MUDr Karel Kameník sro, Brno
  - Kardiologicka ambulance Brno sro, Brno
  - Kardio Elbl sro, Brno
  - Ordinace pro choroby srdce sro, Chomutov
  - Nemocnice Ceske Budejovice as, České Budějovice
  - Dika centrum sro, Havirov - Mesto
  - Kardio Holesov sro, Holešov
  - MUDr Ladislava Harrerova, kardiologicka ordinace, Hradec Králové
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Nemocnice Jihlava po, Jihlava
  - Kardio Michal Cepelak sro, Klatovy IV
  - MUDr Zbynek Kosek, kardiologicka ambulance sro, Mladá Boleslav
  - Edumed sro, Náchod
  - PreventaMed sro, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava
  - Mestska nemocnice Ostrava, po, Ostrava - Moravska Ostrava
  - Pedicor Trial sro, Ostrava-Dubina
  - Nemocnice Pardubickeho kraje as, Pardubice
  - Fakultni nemocnice Plzen, Pilsen
  - Policska nemocnice sro, Polička
  - Ordinace pro choroby srdce a cev, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Institut klinicke a experimentalni mediciny, Prague
  - Milan Kvapil sro, Prague
  - Interni a kardiologicka ordinace, Prague
  - Endokrinologie Cerny Most sro, Prague
  - Kardiologicke centrum MUDr Janky Skrobakove sro, Praha 5 - Smichov
  - Poliklinika Ravak Pribram, Pribram VIII
  - Kardio Vaclavik sro, Interni a kardiologicka ambulance, Přerov
  - Kardiologicka ambulance MUDr Ferkl, sro, Trutnov
  - Clinical Trials Service sro, Uherské Hradiště
  - Cardio Research sro, Zlín
  - Krajska nemocnice T Bati as, Zlín
- Denmark (16):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Aarhus N
  - Rigshospitalet, Copenhagen O
  - Sydvestjysk Sygehus, Esbjerg
  - Sanos Gandrup, Gandrup
  - Herlev Gentofte Hospital, Herlev
  - Sanos Clinic, Herlev
  - Regionshospitalet Gødstrup, Herning
  - Holbaek Sygehus, Holbæk
  - University of Fredriksberg Hospital, København NV
  - Amager Hospital, København S
  - Sjaellands Universitetshospital, Roskilde, Roskilde
  - Slagelse Sygehus, Slagelse
  - Svendborg Sygehus, Svendborg
  - Sanos Vejle, Vejle
  - Regionshospitalet Viborg, Viborg
- Estonia (4):
  - Innomedica, Tallinn
  - Center for Clinical and Basic Research Tallinn, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- Finland (5):
  - Helsinki University Central Hospital, Helsinki
  - Satucon Oy/Kuopion tyoterveys, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Suomen Terveystalo Oy, Turku
- France (19):
  - Centre Hospitalier Regional Universitaire de Besancon, Hopital Jean Minjoz, Besançon
  - Hospices Civils de Lyon Groupement Hospitalier Est, Hopital Louis Pradel, Bron
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital Trousseau, Chambray-lès-Tours
  - Centre Hospitalier Compiegne-Noyon, Compiègne
  - Centre Hospitalier Universitaire de Dijon - Hopital Francois Mitterrand, Dijon
  - Centre Hospitalier Regional Universitaire de Lille - Hopital Claude Huriez, Lille
  - Hopital de la Conception, Marseille
  - Hopital Saint-Joseph, Marseille
  - Centre Hospitalier Universitaire de Montpellier - Hopital Lapeyronie, Montpellier
  - Centre Hospitalier Universitaire de Nantes - Hopital Guillaume et Rene Laennec, Nantes
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur, Nice
  - Hopital Saint Antoine, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Hopital Bichat Claude Bernard, Paris
  - Centre Hospitalier Universitaire de Reims - Hopital Robert Debre, Reims
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Centre Hospitalier Universitaire de Strasbourg - Hopital de Hautepierre, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse - Hopital Rangueil, Toulouse
  - Polyclinique Vauban, Valenciennes
- Germany (30):
  - Universitaetsklinikum Aachen, Aachen
  - Universitaets-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Universitaetsklinikum der Ruhr-Universitaet Bochum, Bad Oeynhausen
  - Velocity Clinical Research GmbH, Berlin
  - Charite - Universitaetsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Charite - Universitaetsmedizin Berlin, Campus Virchow, Berlin
  - Klinikum Links der Weser, Bremen
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Dresden, Dresden
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Frankfurt, Frankfurt am Main
  - ClinPhenomics CVC GmbH, Frankfurt am Main
  - Evangelisches Krankenhaus Goettingen-Weende, Göttingen
  - Universitaetsmedizin Goettingen - Georg-August-Universitaet, Göttingen
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Cardiologicum Hamburg GbR, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - B Braun Ambulantes Herzzentrum Kassel mvz GmbH, Kassel
  - Universitaetsklinikum Leipzig, Leipzig
  - Otto von Guericke Universitaet Magdeburg, Magdeburg
  - Universitaetsklinikum Mannheim, Mannheim
  - Kardiologische Praxis Doktor Jens Taggeselle, Markkleeberg
  - Klinikum rechts der Isar der TUM, München
  - Universitaetsklinikum Muenster, Münster
  - Kardiologische Gemeinschaftspraxis Papenburg, Papenburg
  - Sana-Klinikum Remscheid GmbH, Remscheid
  - Lipidambulanz der Universitaet Rostock, Rostock
  - Klinik am See - Ruedersdorf, Rüdersdorf
  - Hegau-Bodensee-Klinikum Singen, Singen
  - Forschungszentrum Ruhr, Witten
- Greece (13):
  - General Hospital of Athens Evaggelismos, Athens
  - Athens Naval Hospital, Athens
  - General Hospital of Athens Ippokrateio, Athens
  - Laiko General Hospital, Athens
  - Alexandra Hospital, Athens
  - Attikon Hospital, Athens
  - Konstantopoulio - Agia Olga Hospital of Nea Ionia, Athens
  - Hygeia Hospital, Athens
  - Metropolitan Hospital, Athens
  - University Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina, Ioannina
  - General Hospital of Mitilini Vostanio, Mytilene
  - General Hospital of Thessaloniki Ahepa, Thessaloniki
- Hong Kong (2):
  - University of Hong Kong, Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin, New Territories
- Hungary (17):
  - Lausmed Kft, Baja
  - Dr Lakatos Ferenc Private Cardiology Practice, Békéscsaba
  - Budapesti Szent Ferenc Korhaz, Budapest
  - High Tech Medical Kft, Budapest
  - Clinexpert Kft, Budapest
  - Gottsegen Gyorgy Orszagos Kardiovaszkularis Intezet, Budapest
  - Semmelweis Egyetem Varosmajori Sziv es Ergyogyaszati Klinika, Budapest
  - Eszak-Pesti Centrum Korhaz - Honvedkorhaz, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Pharma4 Trial Kft, Gyöngyös
  - BKS Research Kft, Hatvan
  - Selye Janos Korhaz, Komárom
  - Borsod-Abauj-Zemplen Varmegyei Kozponti Korhaz es Egyetemi Oktatokorhaz, Miskolc
  - Dr Nagy Laszlo Kardiologiai maganrendeles es SMO, Orosháza
  - Vita Verum Medical Bt, Székesfehérvár
  - Belvarosi Egeszseghaz Kft, Zalaegerszeg
  - Obudai Egeszsegugyi Centrum Kft, Zalaegerszeg
- Iceland (2):
  - Hjartamidstodin, Kopavogur
  - Thjonustumidstod Rannsoknaverkefna, Kopavogur
- Italy (20):
  - Ospedali dell Ovest Vicentino, Arzignano
  - IRCCS Azienda Ospedaliero Universitaria di Bologna Policlinico di Sant Orsola, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Sant Anna e San Sebastiano, Caserta
  - Azienda Ospedaliera Cannizzaro, Catania
  - Azienda Ospedaliera Universitaria Renato Dulbecco, Catanzaro
  - Azienda Ospedaliera Universitaria di Ferrara Arcispedale Sant Anna, Cona FE
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino IRCCS, Genova
  - IRCCS Centro Cardiologico Monzino, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Ospedale degli Infermi di Rivoli, Rivoli
  - Fondazione Policlinico Tor Vergata, Roma
  - Azienda Ospedaliera Policlinico Umberto I, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano MI
  - Azienda Ospedaliera Universitaria Ospedale San Giovanni di Dio e Ruggi D Aragona, Salerno
  - Multimedica, Sesto San Giovanni (MI)
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
- Japan (65):
  - Kasugai Municipal Hospital, Kasugai-shi, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Tosei General Hospital, Seto-shi, Aichi-ken
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - Hirosaki University Hospital, Hirosaki-shi, Aomori
  - Asahi General Hospital, Asahi-shi, Chiba
  - New Tokyo Heart Clinic, Matsudo-shi, Chiba
  - University of Fukui Hospital, Yoshida-gun, Fukui
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Kokura Memorial Hospital, Kitakyushu-shi, Fukuoka
  - Japan Community Health care Organization Kyushu Hospital, Kitakyushu-shi, Fukuoka
  - Gifu Heart Center, Gifu, Gifu
  - Ogaki Municipal Hospital, Ogaki-shi, Gifu
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima, Hiroshima
  - Asahikawa City Hospital, Asahikawa-shi, Hokkaido
  - Hakodate Municipal Hospital, Hakodate-shi, Hokkaido
  - Tomakomai City Hospital, Tomakomai-shi, Hokkaido
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji-shi, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanazawa Medical University Hospital, Kahoku-gun, Ishikawa-ken
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Iwate Prefectural Central Hospital, Morioka, Iwate
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - Tenyoukai Chuo Clinic, Kagoshima, Kagoshima-ken
  - Fujisawa City Hospital, Fujisawa-shi, Kanagawa
  - Tokai University Hospital, Isehara-shi, Kanagawa
  - Kitasato University Hospital, Sagamihara-shi, Kanagawa
  - Showa University Fujigaoka Hospital, Yokohama, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Yokohama Minami Kyousai Hospital, Yokohama, Kanagawa
  - Yokohama Sakae Kyosai Hospital Federation of National Public Service Personnel Mutual Association, Yokohama, Kanagawa
  - Chikamori Hospital, Kochi, Kochi
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Sendai Cardiovascular Center, Sendai, Miyagi
  - Miyazaki Medical Association Hospital, Miyazaki, Miyazaki
  - Shinshu University Hospital, Matsumoto-shi, Nagano
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Kawasaki Medical School Hospital, Kurashiki-shi, Okayama-ken
  - Rinku General Medical Center, Izumisano, Osaka
  - Sakurabashi Watanabe Advanced Healthcare Hospital, Osaka, Osaka
  - Osaka City General Hospital, Osaka, Osaka
  - Osaka Police Hospital, Osaka, Osaka
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Saga-ken Medical Centre Koseikan, Saga, Saga-ken
  - Ageo Central General Hospital, Ageo-shi, Saitama
  - Sanai Hospital, Saitama-shi, Saitama
  - National Hospital Organization Shizuoka Medical Center, Sunto-gun, Shizuoka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Minamino Cardiovascular Hospital, Hachioji-shi, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo
  - Japanese Red Cross Musashino Hospital, Musashino-shi, Tokyo
  - Ome Medical Center, Ome-shi, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - Tokyo Womens Medical University Hospital, Shinjuku-ku, Tokyo
  - Toyama Prefectural Central Hospital, Toyama, Toyama
  - Seiyu Memorial Hospital, Wakayama, Wakayama
  - Tokuyama Central Hospital, Shunan-shi, Yamaguchi
  - University of Yamanashi Hospital, Chuo-shi, Yamanashi
- Lithuania (6):
  - Klinikiniai sprendimai, Alytus
  - Klinikiniai sprendimai, Kaunas
  - Saules Seimos Medicinos Centras, Kaunas
  - Kardiologijos ir reabilitacijos klinika, Klaipėda
  - Pirmoji viltis JSC, Šiauliai
  - Vilnius University Hospital Santaros Clinic Public Institution, Vilnius
- Mexico (9):
  - Virgen Cardiovascular Research SC, Guadalajara, Jalisco
  - Eukarya PharmaSite, Monterrey, Nuevo León
  - Centro para el Desarrollo de la Medicina y de Asistencia Medica Especializada SC, Culiacán, Sinaloa
  - Consultorio de Medicina Especializada del Sector Privado, Xalapa, Veracruz
  - Centro de investigacion Cardiometabolica, Aguascalientes
  - Fundacion Cardiovascular de Aguascalientes AC, Aguascalientes
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Scientia Investigacion Clinica SC, Chihuahua City
  - Procliniq Investigacion Clinica, Mexico City
- Netherlands (29):
  - Meander Medisch Centrum, Amersfoort
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Rijnstate Ziekenhuis, Arnhem
  - Bravis ziekenhuis, locatie Roosendaal, Bergen op Zoom
  - Amphia ziekenhuis, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Catharina Ziekenhuis, Eindhoven
  - Maxima Medisch Centrum, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - Zuyderland Medisch Centrum, Heerlen
  - Spaarne Gasthuis, locatie Haarlem Zuid, Hoofddorp
  - Dijklander Ziekenhuis Hoorn, Hoorn
  - Leids Universitair Medisch Centrum, Leiden
  - Alrijne Ziekenhuis, Leiderdorp
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - D and A Research and Genetics, Sneek
  - Haaglanden MC, The Hague
  - Haga Ziekenhuis, The Hague
  - Ziekenhuis Rivierenland, Tiel
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
  - Universitair Medisch Centrum Utrecht, Utrecht
  - VieCuri Medisch Centrum, Venlo
- Norway (3):
  - Oslo Universitetssykehus HF Aker sykehus, Oslo
  - Oslo Universitetssykehus HF, Aker sykehus, Oslo
  - Skedsmo Medisinske senter, Skedsmokorset
- Poland (24):
  - American Heart of Poland Spolka Akcyjna, Bełchatów
  - American Heart of Poland Spolka Akcyjna Polsko-Amerykanskie Kliniki Serca, Bielsko-Biala
  - American Heart of Poland Spolka Akcyjna, Chrzanów
  - American Heart of Poland Spolka Akcyjna Polsko-Amerykanskie Kliniki Serca, Dąbrowa Górnicza
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - NZOZ Medica Jerzy Cygler, Giżycko
  - American Heart of Poland Spolka Akcyjna Polsko-Amerykanskie Kliniki Serca, Kędzierzyn-Koźle
  - Jaroslaw Ciosek Rajtar-Medica Centrum Medyczne, Krakow
  - Wojewodzki Specjalistyczny Szpital im dr Wladyslawa Bieganskiego w Lodzi, Lodz
  - Miedziowe Centrum Zdrowia SA, Lubin
  - CenterMed Spzoo Centermed Lublin, Lublin
  - Clinical Best Solutions Sp zoo Spolka Komandytowa Gabinet Lekarski, Lublin
  - NZOZ Twoja Przychodnia Spzoo Twoja Przychodnia Spzoo, Lublin
  - Uniwersyteckie Centrum Stomatologii I Medycyny Specjalistycznej Spolka z ograniczona odpowiedzialnos, Poznan
  - KO-MED Centra Kliniczne Sp zoo KO-MED Centra Kliniczne Pulawy, Puławy
  - American Heart of Poland Spolka Akcyjna Polsko-Amerykanskie Kliniki Serca, Sztum
  - American Heart of Poland Spolka Akcyjna Polsko-Amerykanskie Kliniki Serca, Tychy
  - FutureMeds Warszawa Centrum, Warsaw
  - Szpital Grochowski imienia Doktora medycyny Rafala Masztaka Spzoo, Warsaw
  - Narodowy Instytut Kardiologii Stefana kardynala Wyszynskiego - Panstwowy Instytut Badawczy, Warsaw
  - Futuremeds spolka z ograniczona odpowiedzialnoscia, Wroclaw
  - Slaskie Centrum Chorob Serca w Zabrzu, Zabrze
  - KO-MED Centra Kliniczne Zamosc, Zamość
  - American Heart of Poland Spolka Akcyjna, Zgierz
- Portugal (13):
  - Unidade de Saude Local de Almada-Seixal, EPE - Hospital Garcia de Orta, Almada
  - Unidade Local de Saude de Amadora-Sintra, EPE, Amadora
  - Unidade Local de Saude da Regiao de Aveiro, EPE - Hospital Infante Dom Pedro, Aveiro
  - Unidade Local de Saude de Braga, EPE, Braga
  - Unidade Local de Saude de Lisboa Ocidental, EPE - Hospital de Santa Cruz, Carnaxide
  - Hospital de Cascais, Cascais
  - Unidade Local de Saude de Coimbra, EPE, Coimbra
  - Unidade Local de Saude do Alto Ave, EPE, Guimarães
  - Unidade Local de Saude de Matosinhos, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - Unidade Local de Saude de Santo Antonio, EPE - Hospital de Santo Antonio, Porto
  - Unidade Local de Saude de Entre Douro e Vouga, EPE - Hospital de Sao Sebastiao, Santa Maria da Feira
  - Unidade Local de Saude da Arrabida, EPE - Hospital de Sao Bernardo, Setúbal
  - Unidade Local de Saude de Gaia-Espinho, EPE, Vila Nova de Gaia
- Romania (8):
  - cmi Cardiologie - Dr Mercea Corina Delia, Baia Mare
  - Spitalul Clinic Universitar de Urgenta Elias, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Matcord Biomedica Buzau, Buzău
  - SC Sal Med SRL, Piteşti
  - Cardio Med Medical Center Targu Mures, Târgu Mureş
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
- Slovakia (20):
  - Alian, sro, Bardejov
  - Narodny ustav srdcovych a cievnych chorob, as, Bratislava
  - Kardiovita sro, Bratislava
  - Nemocnica s poliklinikou Brezno, no, Brezno
  - Intergal, sro, Kláštor pod Znievom
  - Medical group Kosice sro, Košice
  - Zarmed, sro, Košice
  - Cardio D and R, sro Kosice, Košice
  - Kardio 1 sro, Lučenec
  - Medi M and M sro, Moldava nad Bodvou
  - Oralek, sro, Námestovo
  - Kardiocentrum Nitra sro, Nitra
  - Kardiomed NZ, sro, Nové Zámky
  - Medikard, sro, Prešov
  - Medispol, sro, Prešov
  - Medilex sro, Rimavská Sobota
  - Tatratrial sro, Rožňava
  - Interna SK, sro, Svidník
  - Areteus sro, Trebišov
  - CardiOr, sro, Trenčín
- South Korea (14):
  - Dong-A University Hospital, Busan
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hospital, Ulsan
  - Yonsei University Wonju Severance Christian Hospital, Wonju-si, Gangwon-do
- Spain (22):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Universitario de Leon, León, Castille and León
  - Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Catalonia
  - Hospital de Sant Joan Despi Moises Broggi, Sant Joan Despí, Catalonia
  - Complexo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Hospital Alvaro Cunqueiro, Vigo, Galicia
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital de Cabueñes, Gijón, Principality of Asturias
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Arnau de Vilanova de Valencia, Valencia, Valencia
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Sweden (7):
  - Falu Lasarett, Falun
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Helsingborgs Lasarett, Helsingborg
  - Clemenstorgets Hjartmottagning, Lund
  - PharmaSite Malmo, Malmo
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Taiwan (9):
  - Hualien Tzu Chi Hospital, Hualien City, Hualien
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Mackay Memorial Hospital Tamsui Branch, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - Veterans General Hospital - Taichung, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District
- United Kingdom (22):
  - Ormeau Clinical Trials Ltd, Belfast
  - Russell Hall Hospital, Birmingham
  - NIHR Patient Recruitment Centre Blackpool, Blackpool
  - NIHR Patient Recruitment Centre Bradford, Bradford
  - West Walk Surgery, Bristol
  - St Richards Hospital, Chichester
  - Rowden Surgery, Chippenham
  - Craigavon Area Hospital, Craigavon
  - Panthera Biopartners - London, Enfield
  - NIHR Patient Recruitment Centre Exeter, Exeter
  - Panthera Biopartners - Glasgow, Glasgow
  - Harefield Hospital, Harefield
  - Wycombe General Hospital, High Wycombe
  - Highlands Clinical Research Facility, Raigmore Hospital, Inverness
  - NIHR Patient Recruitment Centre Leicester, Leicester
  - Lincoln County Hospital, Lincoln
  - Queen Mary University of London, London
  - Hammersmith Hospital, London
  - University Hospital Llandough, Penarth
  - The Adam Practice, Poole
  - Panthera Biopartners - Preston, Preston
  - Lister Hospital, Stevenage

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Byambaa E, Roshanravan B, Berglund L. Lipoprotein(a) and CKD: Insights into New Therapeutic Opportunities. Clin J Am Soc Nephrol. 2025 Dec 2. doi: 10.2215/CJN.0000000968. Online ahead of print. PMID 41329869
- [Derived] Nicholls SJ, Nelson AJ, Michael LF. Oral agents for lowering lipoprotein(a). Curr Opin Lipidol. 2024 Dec 1;35(6):275-280. doi: 10.1097/MOL.0000000000000953. Epub 2024 Sep 25. PMID 39329200
- [Derived] Dimitriadis K, Theofilis P, Iliakis P, Pyrpyris N, Dri E, Sakalidis A, Soulaidopoulos S, Tsioufis P, Fragkoulis C, Chrysohoou C, Tsiachris D, Tsioufis K. Management of dyslipidemia in coronary artery disease: the present and the future. Coron Artery Dis. 2024 Sep 1;35(6):516-524. doi: 10.1097/MCA.0000000000001375. Epub 2024 Apr 29. PMID 38682459
- [Derived] Karp A, Jacobs M, Barris B, Labkowsky A, Frishman WH. Lipoprotein(a): A Review of Risk Factors, Measurements, and Novel Treatment Modalities. Cardiol Rev. 2025 Jul-Aug 01;33(4):352-358. doi: 10.1097/CRD.0000000000000667. Epub 2024 Feb 28. PMID 38415744
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com